CLINICAL TRIAL: NCT03061643
Title: SAMSUNG MEDICAL CENTER
Brief Title: An Open Label Phase II Study of Biweekly Docetaxel Plus Androgen-Deprivation Therapy in Patients With Previously-Untreated, Metastatic, Prostatic Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park, Se-Hoon, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01-005
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Docetaxel PLUS ADT (Experimental): receive docetaxel 40 mg/m2 IV every 2 weeks plus ADT
  Interventions: Drug: Docetaxel; Other: Androgen-Deprivation Therapy (ADT)

INTERVENTIONS:
Drug: Docetaxel — docetaxel 40 mg/m2 IV every 2 weeks plus ADT
Other: Androgen-Deprivation Therapy (ADT) — docetaxel 40 mg/m2 IV every 2 weeks plus ADT

SUMMARY:
Study of Biweekly Docetaxel plus Androgen-Deprivation Therapy (ADT) in Patients with Previously-Untreated, Metastatic, Prostatic Adenocarcinoma

DETAILED DESCRIPTION:
Although surgical or medical castration is considered standard treatment in hormone-naïve PC patients, some patients with extensive metastatic disease, including visceral or bone involvement beyond axial skeleton, have shorter survival. Based on the recent randomized trials (CHAARTED, GETUG-AFU15 and STAMPEDE), hormone-naïve men with metastatic, high-volume PC should be offered docetaxel plus ADT. However, side effects from standard 3-weekly 75 mg/m2 docetaxel can be substantial. In addition, a prospective trial is needed to determine whether early docetaxel chemotherapy in combination with ADT is beneficial in Korean men. Considering our own experiences with docetaxel, a dose intensity of 20 mg/m2/week (equivalent to 60 mg/m2 3-weekly or 40 mg/m2 biweekly) should be tested in the prospective trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male at least 20 years of age.
2. Subject has a histologically or cytologically confirmed diagnosis of adenocarcinoma of prostate.
3. Subject has radiologic and clinical evidence of metastatic disease initially or after treatment for localized disease. They must have metastatic or progressive disease for which there is no further curative treatment available.
4. Subject has an ECOG performance status of 0 to 1.
5. Subject has a life expectancy of 3 months or more.
6. At least 4 weeks since the last surgical procedures or radiotherapy prior to enrolment. Subjects must have recovered to <Grade 2 from all acute toxicities or toxicity must be deemed irreversible by the investigator.
7. Acceptable hematologic status (without growth factor support or transfusion dependency):
8. Acceptable renal function with serum creatinine
9. Acceptable liver function:
10. Subject must agree to use an adequate method of contraception (condom) if he is having sex with a woman of childbearing potential or with a woman who is pregnant.
11. Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

1. Ongoing treatment with an anticancer agent not contemplated in this protocol
2. Pathologic finding consistent with neuroendocrine or small cell carcinoma
3. Any history of clinically relevant coronary artery disease or myocardial infarction within the last 3 years, New York Heart Association (NYHA) grade III or greater congestive heart failure, cerebrovascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
4. Non-tolerable >Grade 2 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1
5. Known uncontrolled brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 4 weeks prior to Cycle 1 Day 1). Subjects that develop brain metastasis during the study may have their treatment interrupted to receive a course of cranial radiation and restart trial medication after a recovery period of at least 1 week. High dose corticosteroids may be employed for the management of cranial radiation but must be tapered off before resuming treatment.
6. Major surgery, other than diagnostic surgery, within 4 weeks prior to Cycle 1 Day 1, without complete recovery.
7. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
8. Subjects who have exhibited allergic reactions to taxanes.
9. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
10. The subject has legal incapacity or limited legal capacity. Dementia or significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Time-to-CRPC (biochemical or clinical) | 24 months

SECONDARY OUTCOMES:
Progression-free survival | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: SEHOON SEHOON, MD,PhD, Principal Investigator — SamsungMedicalCenter
Locations (1):
- Samsung Medical Center, Seoul, South Korea